CLINICAL TRIAL: NCT02609061
Title: Platelet Rich Fibrin Combined With 1% Alendronate Gel in Treatment of Mandibular Degree II Furcation Defects: A Randomized Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin+1% Alendronate in Treatment of Mandibular Degree II Furcation Defects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Dept of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014T
Record Dates: First submitted 2015-11-15; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group 1 (Active Comparator): Scaling and Root Planing (SRP) with Open flap debridement (OFD) alone for treating furcation defect
  Interventions: Procedure: Open flap debridement (OFD)
- Group 2 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF) for treating furcation defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)
- Group 3 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1% Alendronate for treating furcation defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)+1% Alendronate (Drug) in gel form

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Open flap debridement (OFD) alone
  Arms: Group 1
Procedure: OFD with Platelet rich fibrin (PRF) — Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement
  Arms: Group 2
Procedure: OFD with Platelet rich fibrin (PRF)+1% Alendronate (Drug) in gel form — Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1% Alendronate gel placement
  Arms: Group 3

SUMMARY:
The present study was designed to evaluate the combined efficacy of PRF and 1% ALN in the treatment of mandibular degree II furcation defects when compared with PRF and open flap debridement (OFD) alone.

DETAILED DESCRIPTION:
Background: Various regenerative materials have been introduced and tested in the treatment of furcation defects. Platelet-rich fibrin (PRF) is a reservoir of growth factors and cytokines which are the key factors for regeneration of bone and maturation of the soft tissue. Alendronate (ALN), a potent member of bisphosphonate group is known to promote tissue regeneration by inhibiting osteoclastic bone resorption and promoting osteoblastogenesis. The present study was designed to evaluate the combined efficacy of PRF and 1% ALN in the treatment of mandibular degree II furcation defects when compared with PRF and open flap debridement (OFD) alone.

Methods: Seventy two mandibular furcation defects were treated with either OFD alone (Group 1), OFD with PRF (Group 2), and OFD with PRF+1% ALN (Group 3). Clinical parameters; site specific plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), relative vertical attachment level (RVAL) and relative horizontal attachment level (RHAL), intrabony defect depth (IBD) were recorded at baseline before surgery and 9 months post-operatively. Percentage radiographic defect fill was evaluated at baseline and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Presence of buccal Class II furcation defects in endodontically vital, asymptomatic mandibular first and second molars with a radiolucency in the furcation area on an intraoral periapical radiograph with probing depth (PD) ≥ 5mm and horizontal ≥ PD 3mm after phase I therapy i.e, scaling and root planing (SRP);
* No history of antibiotic or periodontal therapy in the preceding 6 months.

Exclusion Criteria:

* Systemic conditions known to affect the periodontal status;
* Medications known to affect the outcomes of periodontal therapy;
* Hematological disorders and insufficient platelet count (<200,000/mm3);
* Pregnancy/lactation;
* Smoking and tobacco use in any form
* Immunocompromised individuals;
* Those having unacceptable oral hygiene (plaque index [PI] >1.5).
* Teeth with furcation involvement, non-vital teeth, and carious teeth indicated for restorations and mobility of at least grade II
* Aggressive periodontitis

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Radiographic bone fill | baseline to 9 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth | baseline to 9 months
  measured in mm
Relative vertical attachment level | baseline to 9 months
  measured in mm
Relative horizontal attachment level | baseline to 9 months
  measured in mm
modified sulcus bleeding index | baseline to 9 months
  0-3 scale
plaque index | baseline to 9 months
  0-3 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Kanoriya D, Pradeep AR, Garg V, Singhal S. Mandibular Degree II Furcation Defects Treatment With Platelet-Rich Fibrin and 1% Alendronate Gel Combination: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Mar;88(3):250-258. doi: 10.1902/jop.2016.160269. Epub 2016 Oct 7. PMID 27712462